CLINICAL TRIAL: NCT05630053
Title: Randomized Controlled Trial to Compare Persona OsseoTi Keel Cementless TKA vs Persona Keel Cemented TKA
Brief Title: Cemented vs Cementless Persona Keel RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMG2022-08K
Record Dates: First submitted 2022-10-18; First posted 2022-11-29 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-03

CONDITIONS: Knee Pain Chronic; Rheumatoid Arthritis; Osteoarthritis; Traumatic Arthritis; Polyarthritis; Avascular Necrosis; Varus Deformity; Valgus Deformity; Flexion Deformity of Knee
Keywords: Total Knee Replacement; Total Knee Arthroplasty; Osteoarthritis; Rheumatoid Arthritis; Cementless; Cementless Knee
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Arthritis; Osteonecrosis

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants should be masked until after the surgical procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Cementless Persona Keel Knee System (Active Comparator): Persona PPS CoCr Cementless Femur and Persona OsseoTi Keel Cementless Tibia
  Interventions: Device: Cementless Persona Knee System
- Cemented Persona Keel Knee System (Active Comparator): Persona Keel Cemented Tibia
  Interventions: Device: Cemented Persona Knee System

INTERVENTIONS:
Device: Cementless Persona Knee System — The Persona Keel Knee system is a total knee system used in the replacement of the knee joint.
  Other Names: Persona PPS CoCr Cementless Femur; Persona PPS Femur; PPS Femur; OsseoTi 0° Spiked Keel Tibia; OsseoTi Tibia; OsseoTi Spiked Keel Tibia; Spiked Keel Tibia; Cementless Tibia
  Arms: Cementless Persona Keel Knee System
Device: Cemented Persona Knee System — The Persona Keel Knee system is a total knee system used in the replacement of the knee joint.
  Other Names: Persona Keel Cemented Tibia; Keel Tibia
  Arms: Cemented Persona Keel Knee System

SUMMARY:
The main objective of this study is to evaluate the safety, performance, and clinical benefits of the Persona Keel cementless and cemented knee.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized controlled trial to demonstrate safety, performance, and clinical benefits of the Persona Keel CR Knee System and instrumentation. Participants that meet eligibility criteria and sign an institutional review board (IRB) Informed Consent form will be randomized to receive either the Persona OsseoTi Keel Cementless System or the Persona Keel Cemented System. Participants will be blinded to which arm they have been randomized to until after surgery.

All study participants will undergo preoperative clinical evaluations prior to their total knee arthroplasty. Investigators will collect clinical data for up to 5 years; follow-up clinic visits will occur at 3 months, 1 year, 2 years, and 5 years after surgery.

A maximum of 10 sites will contribute to this study. There will be a maximum of 300 participants enrolled (150 Cementless, 150 Cemented).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is of legal age and skeletally mature
2. Patient is willing and able to provide written Informed Consent by signing and dating the IRB/EC approved Informed Consent document
3. Patient is willing and able to complete scheduled follow-up evaluations as defined in the study protocol
4. Independent of study participation, patient qualifies for either cemented or cementless total knee arthroplasty based upon physical exam and medical history, and meets the approved indications for use of the commercially available Persona Keel Knee System with appropriately matched Zimmer Biomet components implanted in accordance with product labeling.

Exclusion Criteria:

1. Patient is unwilling to sign the Informed Consent
2. Patient is currently participating in any other surgical intervention or pain management study
3. Patient is pregnant or considered a member of a protected (vulnerable) population whose inclusion in the study would be inappropriate (e.g., prisoner; pediatric patients)
4. Patient has a mental or neurologic condition who is unwilling or incapable of following postoperative care instructions
5. Patient has a condition which would, in the judgement of the Investigator, place the patient at undue risk or interfere with the conduct of the study
6. Patient is institutionalized or is a known drug abuser, a known alcoholic or cannot understand the requirements of study participation
7. Patient is scheduled to undergo simultaneous bilateral total knee arthroplasty

   Study Device-Specific Exclusion Criteria:
8. Previous history of infection in the affected joint and/or other local/systematic infection that may affect the prosthetic joint
9. Insufficient bone stock on femoral or tibial surfaces.
10. Neuropathic arthropathy
11. Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
12. A stable, painless arthrodesis in a satisfactory functional position
13. Severe instability secondary to the absence of collateral ligament integrity
14. Rheumatoid arthritis (RA) accompanied by an ulcer of the skin or a history of recurrent breakdown of the skin
15. The kinematic alignment surgical technique is contraindicated for patients with greater than 5° valgus deformity with MCL insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2032-05 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Oxford Knee Score (OKS) | 5 years
  A 12-item PROM was specifically designed and developed to assess function and pain after TKA. This tool is short, reproducible, valid, and sensitive to clinically important changes. Possible scores range from a minimum 0 to maximum 48 points, with higher scores indicating less pain and fewer functional limitations. The primary endpoint is based on the change in OKS scores from baseline to 2-year postoperative follow-up as well as from baseline to 5-year postoperative follow-up.

SECONDARY OUTCOMES:
Survival Rate of Implant | 5 years
  Survival Rate (Survivorship) will be both assessed by revision/additional surgeries to the affected joint due to aseptic loosening only or by revision, removal, exchange of the implanted device due to any reason. Aseptic loosening and other reasons for additional surgeries may be identified by radiographic imaging.
Frequency and types of Adverse Events | 5 years
  The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.
EuroQol-5 Dimension-5 Level (EQ-5D-5L) Questionnaire | 5 years
  The EQ-5D-5L instrument comprises a short descriptive system questionnaire and a visual analogue scale (EQ VAS). The questionnaire produces an "index" score that ranges from 0 to 1, where 0 is the value of a health state equivalent to dead; and 1 is the value of full health, with higher scores indicating higher health utility.
  The EQ VAS is a 0 -100 scale where patients are asked to indicate their overall health on the day of questionnaire completion. 100 indicates the best health imaginable and 0 indicates the worst health imaginable.
  Change in Index and EQ VAS scores will be compared from baseline to 2-year follow-up as well as from baseline to 5-year postoperative follow-up for each cohort (cemented or cementless). This change will also be compared between the cohorts (delta from baseline to 2 years and baseline to 5 years in the cementless group compared to the same delta in the cemented group).
Numeric Rating Scale (Pain) | 5 years
  The 11-item pain NRS asks patients to rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"). It is the most widely used instrument for pain screening with higher scores indicating greater pain intensity.
Patient Expectations Pre- and Post-op | 5 years
  Per the 2011 Knee Society scoring manual: "[This] is a three-question fifteen-point scale that is collected pre-operatively and post-operatively. The pre-operative questions reflect the patient's opinion on the extent to which the patient expects that the operation will improve their knee pain, and their ability to perform their activities of daily living and recreational activities.
  The post-operative questions reflect the extent to which the outcome after the operation has met the patient's pre-operative expectations with respect to pain and function."
  Higher scores preoperatively indicate more positive expectations of the patient's total knee replacement surgery, and higher scores postoperatively indicate
Rate of Radiolucencies | 5 years
  Radiographic parameters to be evaluated include, but are not limited to, radiolucencies, osteolysis, hypertrophy, subsidence, and heterotopic ossification. All radiographic evaluations performed according to the protocol will be reviewed by the investigator at the time of the evaluation for significant radiographic findings.

OTHER OUTCOMES:
Operative Room Time | During surgery
  Evaluation of differences in operative times between implantation of cemented and cementless systems.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Centura Health, Westminster, Colorado
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Oregon Health & Science University, Portland, Oregon
  - Rothman Institute, Bryn Mawr, Pennsylvania
  - Lehigh Valley Hospital - Dickson City, Dickson City, Pennsylvania
  - Houston Methodist Hospital, Houston, Texas
  - Anderson Orthopaedic Research Institute, Alexandria, Virginia